CLINICAL TRIAL: NCT06032676
Title: Surgical Decision Making in Necrotising Enterocolitis - a Prospective Qualitative Study of Surgeons
Brief Title: Qualitative Study of Surgeons With Prospective Patient Follow-up
Acronym: NECqual
Status: Recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM CHI1209; NIHR (Other Grant/Funding Number: NIHR302541)
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Necrotizing Enterocolitis
Keywords: surgical decision making; neonatology; qualitative research; Necrotising enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants with necrotising enterocolitis reviewed by a surgeon: Infant with suspected or confirmed NEC undergoing review by surgeon, regardless of outcome of that review (i.e. surgery indicated or not)

SUMMARY:
Necrotising enterocolitis (NEC) is a devastating disease which causes severe bowel inflammation resulting in babies becoming critically unwell. It mainly affects premature babies (who can be born as early as 22 weeks) in the first few weeks of life. A quarter of babies don't respond to intensive care treatment and require surgery to remove bowel which has died to prevent them from getting sicker. Sadly, about a third of the most unwell babies don't survive and those that do have a high incidence of significant long-term health problems.

Deciding which babies will benefit from surgery is challenging and there are no objective methods used to do this currently. Surgeons must weigh up the risks and benefits of performing major surgery on a tiny baby in the knowledge that surgery itself may cause harm. This uncertainty causes delays in performing surgery. Those that have a delay are more likely to have a poor outcome.

In order to improve these unfavourable outcomes it is essential to understand and define current practice in detail (i.e. indications and timing for surgery) and understand how this may be associated with outcome. These outcomes are both short term, including mortality and ability to tolerate enteral nutrition, and long term which include neurodevelopmental outcomes at 2 years of life.

To do this the investigators will undertake a multicentre mixed methods study with qualitative interview of consultant paediatric surgeons shortly after making a decision to operate, or not, on a baby with NEC. The investigators will then take consent from the parents/guardian of the infant to follow-up their clinical outcomes using data linkage to routinely collected data, within the national neonatal research database. Outcomes of interest include survival, feeding outcomes, further surgical procedures and neurodevelopment at 2 years.

DETAILED DESCRIPTION:
Necrotising enterocolitis (NEC) predominately affects pre-term infants and consists of a severe bowel inflammation which can lead to necrosis. The number of babies at highest risk of developing NEC is rising as survival of extremely preterm babies improves. Whilst unanswered questions remain regarding the aetiology of NEC, the clinical presentation is that of an acutely unwell baby, with abdominal distension requiring intensive care support due to activation of a systemic inflammatory response.

About a quarter of babies will require surgery due to bowel perforation, suspected necrotic bowel or failure to improve with intensive care treatment alone. Most commonly, ischaemic, non-viable gut is found at laparotomy and hence removed. In 1-in-20 surgical procedures the extent of the non-viable gut is so great that survival is not possible.

Surgical practice, including decision-making, in NEC has been previously shown to vary from surgeon to surgeon with no set criteria for when an infant is no longer responding to medical treatment and should have surgery. It can be particularly challenging given that babies with the disease are of extreme prematurity and some weigh as little as 500 grams. There is a real risk of causing harm during surgery hence it is essential that the benefits outweigh the risk. Unfortunately short and long-term outcomes for surgical NEC are poor including mortality in 35% following surgery and 59% of survivors experience neurodevelopmental problems. Recent evidence suggests that earlier surgery for NEC is beneficial and is associated with better outcomes than delayed surgery. Additionally, 20% of neonates with NEC die before surgery which is potentially avoidable with more effective identification of the need for surgery.

In order to improve these unfavourable outcomes it is essential to understand and define current practice in detail (i.e. indications and timing for surgery) and understand how this may be associated with outcome. These outcomes are both short term, including mortality and ability to tolerate enteral nutrition, and long term which include neurodevelopmental outcomes at 2 years of life.

This prospective mixed methods study is entirely observation and involves no intervention. Inclusion in the study is on the basis of fully informed consent.

Study flow is as follows:

1. Initial surgeon interview - After the site setup, all consultant paediatric surgeons that treat infants with NEC will be invited to participate and provided with a participant information sheet along with a consent form. A baseline interview will be conducted with each participating surgeon via telephone based on hypothetical patients. The interview will follow a semi-structured guide. The interview will be recorded for transcription purposes. Thematic analysis will then be undertaken.
2. Clinical Review of Infants with NEC by Consultant Surgeon - Infants will be eligible for inclusion if they have confirmed NEC or their most likely diagnosis is NEC, and are reviewed by a consultant surgeon for consideration of surgery at a study site. The local clinical team or research team will notify the study coordinator that this review has taken place.
3. Qualitative surgeon interview about Review and Decision to Operate or Not - Qualitative interviews will be conducted via telephone as soon as possible after the clinical review by the surgeon. Interviews will be semi-structured, lasting approximately 10 minutes, and follow a topic guide. The interview will be recorded for transcription purposes. Thematic analysis will then be undertaken.
4. Parent Consent and Data Collection - Following the qualitative interview of the surgeon, the parents of the infant who underwent clinical review will be approached for consent to record their infant's details and parental contact information. This process will occur prior to hospital discharge. Data will be collected to allow linkage to the National Neonatal Research Database (NNRD) which routinely collects data on infants admitted to neonatal units nationally.
5. Initial Follow-up - 52 Weeks Corrected Gestational Age - Seven months after the end of data collection (1st May 2025), a list of patients using BadgerNet numbers and dates of birth, will be securely sent to the National Neonatal Research Database (NNRD) via NHS.net email in order to identify the infants on the NNRD. The requested data for each infant will be censored at 52 weeks corrected gestational age. The analysis will focus on identifying associations between the thematic interview analysis and the outcomes of the infants. These groups based on outcome are:

   * Survival and non survival
   * Survival and non-survival or parental nutrition dependence at discharge
   * Surgery after initial surgical review and continued medical management
6. Further Follow-up - 2 Years of Age - the NNRD will be interrogated again on 1st January 2027 using the same procedures used during the initial follow-up. Additional outcomes of interest at this stage are two year outcome assessment date, developmental outcomes and cerebral palsy diagnosis. Associations between these outcomes and themes identified during surgeon interview will again be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Infant with suspected or confirmed NEC undergoing review by surgeon, regardless of outcome of that review (I.e. surgery indicated or not).

   Exclusion Criteria:
2. Lack of consent from surgeon to undertake interview.
3. Lack of consent from parents to follow-up outcomes of infant.

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infant with necrotising enterocolitis undergoing review by paediatric surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | At 52 weeks corrected gestational age and at 2 years age.
  Mortality

SECONDARY OUTCOMES:
Death or parental nutrition dependence | Hospital discharge (up to 52 weeks corrected gestational age)
  Death or parental nutrition dependence versus survivors not requiring parental nutrition

CONTACTS AND LOCATIONS:
Overall Officials: Nigel J Hall, Principal Investigator — University of Southampton
Locations (1):
- University Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data available by reasonable request at end of study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From October 2028 for 10 years.
Access Criteria: Researchers by reasonable request to PI.